CLINICAL TRIAL: NCT01421836
Title: Prospective Study Comparing EUS Guided Biliary Drainage and ERCP With Stent Placement for Malignant Biliary Obstruction
Brief Title: Prospective Study Comparing EUS vs ERCP Stent Insertion for Malignant Biliary Obstruction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Hyuck Lee, Professor of Department of Medicine,Samsung Medical Center,Sungkyunkwan University School of Medicine, Samsung Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-03-101-001
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Tumor Appearance of Biliary System Obstruction
Keywords: stent patency; EUS guided insertion; ERCP guided insertion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERCP guided stent insertion (Active Comparator)
  Interventions: Procedure: ERCP-guided stent insertion
- EUS guided stent insertion (Active Comparator)
  Interventions: Procedure: EUS guided stent insertion

INTERVENTIONS:
Procedure: ERCP-guided stent insertion — ERCP guided stent insertion for malignant biliary obstruction
  Other Names: ERCP-guided metal stent insertion
  Arms: ERCP guided stent insertion
Procedure: EUS guided stent insertion — EUS-guided stent insertion for malignant biliary obstruction
  Other Names: EUS-guided metal stent insertion
  Arms: EUS guided stent insertion

SUMMARY:
1. Purpose of the study

   -To compare stent patency and complication rate between endoscopic ultrasound (EUS) guided stent insertion and endoscopic retrograde cholangiopancreatography (ERCP) guided stent insertion for malignant biliary obstruction
2. Subjects of the study

   -Patients who have biliary obstruction owing to malignant tumors
3. Methods of the study

   * Prospective randomized controlled study
   * Patients were enrolled randomly in two groups, EUS guided stent insertion group or ERCP guided stent insertion group
   * Patients will get assigned procedure (EUS guided stent insertion or ERCP guided stent insertion)for decompression of malignant biliary obstruction
   * After the procedure, regular follow up, blood test,and imaging test will be done to check sufficient biliary decompression,stent patency and complications.

DETAILED DESCRIPTION:
1. Inclusion criteria 1) age: 18 - 80 2) a patients who had common bile duct dilatation because of malignant distal common bile duct obstruction in radiologically 3) Hyperbilirubinemia (total bilirubin >= 1.5 mg/dl) 4) inoperable state 5) a patients who agree to join this study
2. Exclusion criteria 1) a patients who can not endure sedation 2) a patients with bleeding tendency (PT > 1.5 INR, PLT < 50,000) 3) a patients with systemic infection 4) a patients who had hilar obstruction

ELIGIBILITY:
Inclusion Criteria:

* distal biliary obstruction due to malignant tumor
* unresectable tumor
* Jaundice

Exclusion Criteria:

* Children
* Hilar obstruction
* Active infection
* Bleeding tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
stent patency (days) | six months

SECONDARY OUTCOMES:
complication rate | six months

CONTACTS AND LOCATIONS:
Overall Officials: Kwanghyuck Lee, MD, phD, Study Director — Division of Gastroenterology, Department of Internal Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, Irwon-dong, Gangnam-gu, South Korea

REFERENCES:
- [Derived] Park JK, Woo YS, Noh DH, Yang JI, Bae SY, Yun HS, Lee JK, Lee KT, Lee KH. Efficacy of EUS-guided and ERCP-guided biliary drainage for malignant biliary obstruction: prospective randomized controlled study. Gastrointest Endosc. 2018 Aug;88(2):277-282. doi: 10.1016/j.gie.2018.03.015. Epub 2018 Mar 30. PMID 29605722